CLINICAL TRIAL: NCT00613210
Title: Sonographic Prediction of Preterm Delivery Between 24-34 Weeks of Gestation
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Limor Man, soroka medical center
Other Study IDs: SOR463907CTIL; 4639
Record Dates: First submitted 2008-01-22; First posted 2008-02-12 (Estimated); Last update posted 2008-02-12 (Estimated); Status verified 2008-01

CONDITIONS: Healthy
Keywords: preterm delivery; shory cervix; amniotic fluid sludge; uterine artery doppler; singeltone; normal amniotic fluid index; without rupter of membranes; 24-34 weeks of gestation
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: None Retained — sonographic measurments

GROUPS / COHORTS (3):
- 1: women without contraction at 24-34 weeks of gestation
- 2: women without contractions between 24-34 weeks of gestation with a history of preterm labor
- 3: women with preterm contractions 24-34 weeks of gestation

SUMMARY:
to evaluate if sonographic measure of short uterin cervix, sludge in amniotic fluid and abnormal doppler of the uterin artery can predict preterm labor

ELIGIBILITY:
Inclusion Criteria:

* pregnancy between 24-34 wees of gestation

Exclusion Criteria:

* lack prenatal care
* fetal malformations stractural or genetical
* plcenta previa
* cerclage
* women who underwent conization of cervix
* polyhydramnious
* premature rupture of membranes
* induction of labor d/t medical condition preterm
* women with hypertension, diabetis or preeclampsia
* susp IUGR
* women with a chronic illness that may interupt pregnancy

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: women that visit a tetriary hospital for follow up
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2008-01; Primary Completion 2008-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Limor Man, Principal Investigator — soroka medical center sonar unit of obstetrics and gynecology department; limor man, MD, Principal Investigator — Soroka University Medical Center